CLINICAL TRIAL: NCT00387829
Title: Randomized Controlled Trial of DuraGen Plus® Adhesion Barrier Matrix to Minimize Adhesions Following Lumbar Discectomy
Brief Title: DuraGen Plus® Adhesion Barrier for Use in Spinal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor voluntarily terminated study
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DURA-US-2006-1
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Spinal Injuries; Adhesions
MeSH Terms: conditions — Spinal Injuries; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Use of DuraGen Plus Adhesion Barrier Matrix as an adhesion barrier in the spine
  Interventions: Device: DuraGen Plus Adhesion Barrier Matrix
- 2 (No Intervention): Control arm is surgery alone (no adhesion barrier)

INTERVENTIONS:
Device: DuraGen Plus Adhesion Barrier Matrix — Application of DuraGen Plus Adhesion Barrier Matrix in spine surgery
  Arms: 1

SUMMARY:
To evaluate the safety and effectiveness of DuraGen Plus® Adhesion Barrier Matrix as an adhesion barrier in spinal surgery to reduce the extent of peridural fibrosis formation and radicular pain in comparison to a control group receiving standard care.

DETAILED DESCRIPTION:
For more information, please visit www.DuragenStudy.com

ELIGIBILITY:
Inclusion Criteria (Abstracted from clinical protocol):

* Patients with radicular pain requiring single-level, lumbar hemi-laminectomy or hemilaminotomy procedures with discectomy in the lower lumbar spine
* Require initial open lumbar surgery for extruded, prolapsed or bulging intervertebral discs
* Requires removal of herniated disc fragment

Exclusion Criteria (Abstracted from clinical protocol):

* Current or historic open traumatic injury to the spine
* Any previous surgery to the lumbar spine or percutaneous tissue destruction or ablation procedures
* Women who are nursing, women who are pregnant and women who are planning to become pregnant during the time of the study
* Any spinal conditions or systemic diseases that would preclude the patient from participation in the clinical trial
* Clinically significant structural disorders
* Known positive for HIV
* Insulin-dependent Diabetes Mellitus patients
* Morbid obesity (Body Mass Index greater than or equal to 40 kg/m2)
* History of alcohol or drug abuse within 2 years prior to randomization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2006-10; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Benzel, MD, Principal Investigator — The Cleveland Clinic Spine Institute
Locations (36):
- United States (36):
  - Ronderos Neurosurgery Center, Providence Hospital, Mobile, Alabama
  - Spine Source, Beverly Hills, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mission Hospital, Mission Viejo, California
  - University of California, San Diego, San Diego, California
  - Spine Institute, Santa Monica, California
  - Southern California Orthopedic Institute, Van Nuys, California
  - Greenwich Neurosurgery/Greenwich Hospital, Greenwich, Connecticut
  - Orthopaedic Specialties Spine Center, Clearwater, Florida
  - The Back Center, Melbourne, Florida
  - University of Miami, Miami, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - University of South Florida, Tampa, Florida
  - Southeastern Orthopedic Center, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - Chicago Institute of Neurosurgery and Neuroresearch, Chicago, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Bluegrass Orthopedics, Lexington, Kentucky
  - Interactive Neuroscience Center, Shreveport, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Columbia Orthopedic Group, Columbia, Missouri
  - Montana Neuroscience Institute Foundation, Missoula, Montana
  - William S. Muir, MD, PC, Las Vegas, Nevada
  - University of Medicine and Dentistry of New Jersey, New Brunswick, New Jersey
  - University of Cincinnati Medical Center / Mayfield Clinic, Cincinnati, Ohio
  - The Cleveland Clinic Spine Institute, Cleveland, Ohio
  - Central Ohio Neurological Surgery, Westerville, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Princeton Brain and Spine Care, Langhorne, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Roger Williams Hospital, Providence, Rhode Island
  - Texas Back Institute, Plano, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Orthopedics Intl., Seattle, Washington
  - Swedish Neuroscience Institute, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 343 patients were randomized in the study (Intent-to-treat population). Four patients received treatment (1 Duragen Plus; 3 Surgery alone), but were not randomized correctly, and were followed-up for safety only. Hence the total patients in the Safety Population is 347.
Groups:
- 1- DuraGen Plus During Surgery: Use of DuraGen Plus Adhesion Barrier Matrix as an adhesion barrier in the spine
- 2 - Surgery Alone: Control arm is surgery alone (no adhesion barrier)
Period: Safety Population
Arm/Group | 1- DuraGen Plus During Surgery | 2 - Surgery Alone
Started | 178 | 169
Completed | 139 | 136
Not Completed | 39 | 33
Period: Intent-to-treat Population
Arm/Group | 1- DuraGen Plus During Surgery | 2 - Surgery Alone
Started | 177 | 166
Completed | 139 | 136
Not Completed | 38 | 30

BASELINE CHARACTERISTICS:
Population: A total of 343 patients were randomized in the study (Intent-to-treat population). Four patients received treatment (1 Duragen Plus; 3 Surgery alone), but were not randomized correctly, and were followed-up for safety only. Hence the total patients in the Safety Population is 347.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1- DuraGen Plus During Surgery | 2 - Surgery Alone | Total
Number analyzed (Participants) | 177 | 166 | 343
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 171 | 162 | 333
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (11.38) | 43.3 (11.27) | 43.0 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 74 | 150
  Male | 101 | 92 | 193
Region of Enrollment [Number; unit: participants]
  United States | 177 | 166 | 343

OUTCOME MEASURES:

1. Primary Outcome: Radiological, Pain, and Functional Outcome Assessments
Description: Radiological score (MRI Outcome score): MRI peridural fibrosis in 5 consecutive 2-D axial Spin Echo T1 axial slices. Score consists of the ratio of total available space in each image and the amount of scar identified (percentage).
  Pain (VAS): Visual Analog Score used to rate the subject's pain.VAS scale is a 100 mm horizontal line, where the far left side of the scale equals (0) no pain and the far right side of the scale (100) equals the worst possible pain.
  Functional outcome score (ODI): Used to assess the effect leg or back pain on everyday life. Questions relate to areas such as walking, lifting, sitting, ability to travel as well as other common activities. Ten questions with scores from 0-5. Calculated as percentage: (Actual score /Maximum overall score (worst disability))*100.
Time Frame: 6 months
Population: Data reported for patients evaluable at 6 months.
Measure: Least Squares Mean (Standard Error); unit: Outcome scores
Arm/Group | 1- DuraGen Plus During Surgery | 2 - Surgery Alone
Number analyzed (Participants) | 147 | 136
Outcome scores
  MRI Outcome Score | 12.375 (0.499) | 12.578 (0.517)
  ODI Score | 6.974 (0.629) | 7.118 (0.639)
  VAS Score | 14.010 (1.610) | 16.696 (1.646)

2. Secondary Outcome: Radiological, Pain, and Functional Outcome Assessments
Description: as for outcome 1
Time Frame: 12 months
Population: Data reported for patients evaluable at 12 months.
Measure: Least Squares Mean (Standard Error); unit: Outcome scores
Arm/Group | 1- DuraGen Plus During Surgery | 2 - Surgery Alone
Number analyzed (Participants) | 133 | 127
Outcome scores
  MRI Outcome Score | 10.046 (0.519) | 9.788 (0.534)
  ODI Score | 6.048 (0.625) | 6.890 (0.633)
  VAS Score | 12.926 (1.612) | 14.378 (1.633)

ADVERSE EVENTS:
Arm/Group | 1- DuraGen Plus During Surgery | 2 - Surgery Alone
Serious Adverse Events (participants affected / at risk) | 18/178 | 19/169
Other Adverse Events (participants affected / at risk) | 100/178 | 106/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1- DuraGen Plus During Surgery (N=178) | 2 - Surgery Alone (N=169)
Inververtebral disc protrusion (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (9)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Faeces Discouloured (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intracranial hypotension (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cervial spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Post laminectomy syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Unirary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Leriche syndrome (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1- DuraGen Plus During Surgery (N=178) | 2 - Surgery Alone (N=169)
Procedural pain (Injury, poisoning and procedural complications) | 5 (8) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 33 (35) | 36 (43)
Inververtebral disc protrusion (Musculoskeletal and connective tissue disorders) | 16 (16) | 13 (13)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 7 (7) | 12 (12)
Pain in extremety (Musculoskeletal and connective tissue disorders) | 17 (20) | 16 (23)
Headache (Nervous system disorders) | 4 (5) | 7 (9)
Hypoaesthesia (Nervous system disorders) | 7 (7) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days